CLINICAL TRIAL: NCT01724736
Title: A Pilot Study to Determine the Effect of a Cobiotic Formulation on the Fecal Bacteroidetes: Firmicutes Ratio in Pre-Diabetic Subjects.
Brief Title: A Pilot Study to Determine the Effect of a Cobiotic Formulation on the Gastrointestinal Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NuMe Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PrCo Study
Record Dates: First submitted 2012-11-06; First posted 2012-11-12 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Pre Diabetic
Keywords: microbiome; prebiotic; cobiotic; NM504; GI microbiome
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Comparator: (Placebo Comparator): Celluose 10g - Matches the total dietary fiber content of NM504 as well as the color and taste. Subjects take 1 dose within 1h prior to either breakfast or lunch and a 2nd dose within 1h prior to the evening meal for 4 weeks.
  Interventions: Drug: Placebo; Drug: NM504:
- NM504: (Active Comparator): Cobiotic formula of GRAS ingredients with a total dietary fiber content of 10g. Subjects take 1 dose within 1h prior to either breakfast or lunch and a 2nd dose within 1h prior to the evening meal for 4 weeks.
  Interventions: Drug: Placebo; Drug: NM504:

INTERVENTIONS:
Drug: Placebo — Celluose 10g - Matches the total dietary fiber content of NM504 as well as the color and taste. Subjects take 1 dose within 1h prior to either breakfast or lunch and a 2nd dose within 1h prior to the evening meal for 4 weeks.
Drug: NM504: — Cobiotic formula of GRAS ingredients with a total dietary fiber content of 10g. Subjects take 1 dose within 1h prior to either breakfast or lunch and a 2nd dose within 1h prior to the evening meal for 4 weeks.

SUMMARY:
This study aims to investigate the effect of a cobiotic formulation, prepared as a smoothie beverage, on the ratio of intestinal microbiota of the Bacteroidetes phylum to those of the Firmicutes phylum in the stool as well as the effect on insulin resistance, gut hormones (PYY) Peptide YY and (GLP-1) Glucagon-like Peptide, ghrelin with perceptions of appetite and satiety.

DETAILED DESCRIPTION:
Human gut microbiome appears to be involved in the regulation of metabolic processes, including digested food components, absorption of fat, metabolism of drugs, and conversion of indigestible foods or partially digested food ingredients to molecules that may signal physiological host mechanisms. The gut microbiome is a complex ecosystem of liquor or chime and microbiota. A change in that habitat may result in microbiota community shifts and consequential changes in brain-gut regulatory interactions. NM504 is a cobiotic formulation composed of 3 (generally recognized as safe; GRAS) food ingredients. One ingredient is a conventional prebiotic fiber. A second ingredient can be fermented but it also is included to change the viscosity of the biome while protecting the mucosal barrier. The 3rd ingredient is an antioxidant with poor bioavailability that alters the redox potential of the biome, selecting for some and against other microbiota growth. In a placebo-controlled double-blinded intervention this trial will investigate the effect of NM504 on the intestinal microbiota as well as markers of glucose regulation in 20 prediabetic adults. The intervention periods last 28 days. Examination of participants will happen at the beginning, weekly and at the end of intervention and will contain anthropometry; blood samples; fecal samples; oral glucose tolerance test; meal tolerance test; and scales to assess appetite, hunger, mood, and bowel habits.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female.
* Stable body weight.
* Stable body weight (+ 11 pounds) in the 3 months prior to the study. Between 18 and 70 years of age, inclusive.
* BMI between 25 and 45 Kg/m2, inclusive. BMI is a measure of your height to weight ratio. (Body Mass Index).
* Fasting blood glucose between 100 and 200 mg/dL, inclusive.

Exclusion Criteria:

* Pregnant or nursing.
* Diabetes or diseases of the liver, pancreas or gastrointestinal tract (except surgery like cholecystectomy, appendectomy or hiatus hernia repair).
* Taking a medication for diabetes, or a medication like systemic glucocorticoids that can affect blood insulin, or a mediation like atypical antipsychotics that alters affect blood sugar or blood insulin, or a medication like atypical antipsychotics that alters body weight, or a medication like antibiotics that can change intestinal bacterial flora, or a medication that alters blood lipids.
* Past history of Bariatric surgery.
* Chronic use of proton pump inhibitors or bulk laxatives.
* Active dependence on alcohol (>14 drinks/week) or illegal drugs.
* following a weight loss regimen.
* Body weight over 350 pounds (.160 kg).
* Any chronic medication [for example: for treatment of conditions like hypothyroidism (like thyroxine), gout (like allopurinol) or hypertension (like propranolol)] that has not had a stable dose for 1 month or longer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in the ratio of Bacteroidetes to Firmicuites ratio in the stool comparing the baseline value to the completion of study value. | 4 weeks
  Abundance of 11 different genera that are characterized in lean and obese individuals will be quantitated and the ratio of abundance of those in the Bacteriodetes phylum to Firmicutes phylum will calculated.

SECONDARY OUTCOMES:
Insulin sensitivity based on homeostasis model assessment (HOMA) | 4 weeks
  Fasting blood glucose and insulin levels will be used to calculate HOMA-IR (insulin resistance) and to estimate insulin sensitivity at baseline and at the completion of the study.
Fasting blood glucose | Weekly for 4 weeks
  Weekly measurements of fasting blood glucose and serum insulin will be performed.
Body weight | Weekly for 4 weeks
  Body weight will be monitored weekly.
Hunger perception | Weekly for 4 weeks
  Visual analog scales to assess appetite and satiety will be used at weekly visits.
Meal tolerance test | 3 weeks
  A fixed meal will be consumed at 3 weeks. Visual analog scales (VAS) for appetite will be used to measure hunger before the meal. A VAS to assess satiety will be used at completion of the meal. Plasma ghrelin, PYY, GLP-1, glucose and insulin will be measured both before the meal and at 1 hour after consumption.
Clinical Chemistry | 4 weeks
  Blood will be obtained at baseline and after 4-weeks of treatment to measure lipids, high-sensitivity C-reactive protein (hsCRP) and glycosylated hemoglobin (HgbA1c).
Fecal profiling | 4 weeks
  Feces will be collected at baseline and after 4 weeks to measure pH, short chain fatty acids, pathogens, branched chain fatty acids and triglycerides to assess changes in the GI microbiome.
Insulin sensitivity based on Oral Glucose Tolerance Testing | 4 weeks
  An oral glucose tolerance test will be performed at baseline and at the completion of the study to estimate insulin sensitivity.
Mood | 4 weeks
  A standardized mood instrument will be used at baseline and at 4 weeks.
Gastrointestinal Symptoms | 4 weeks
  A survey to measure GI symptoms, changes in bowel habits and changes in stool characteristics will be performed on weekly visits for 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States